CLINICAL TRIAL: NCT07353320
Title: Effects of Probiotics on Alleviating Anxiety and Depression and Gut Microbiota
Brief Title: Probiotics Regulate Intestinal Health and Alleviate Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20251224
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-04

CONDITIONS: Anxiety Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : probiotics group (Experimental): 5 billion CFU/day BC99 and protein powder; Storage: sealed, protected from light, placed in a cool and dry place.
  Interventions: Dietary Supplement: probiotics group
- Placebo Comparator : placebo group (Placebo Comparator): Dextrin powder, 1 bags per day; Storage: sealed, protected from light, placed in a cool and dry place.
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: probiotics group — The intervention lasted 8 weeks, with follow-ups at weeks 0 and 12.
  Arms: Experimental : probiotics group
Dietary Supplement: Placebo Group — The intervention lasted 8 weeks, with follow-ups at weeks 0 and 12.
  Arms: Placebo Comparator : placebo group

SUMMARY:
This study is a randomized, double-blind, placebo-controlled trial aimed primarily at investigating the effects of Weizmannia coagulans BC99 on alleviating anxiety and depression and the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-65 years.
2. Individuals experiencing scientific research, employment-related, or occupational stress, including graduate students or community-dwelling adults with job-related pressure.
3. A Hamilton Depression Rating Scale (HAMD-17) score ≥ 8 and/or a Hamilton 4) Anxiety Rating Scale (HAMA-14) score ≥ 7 at screening.

5)Ability and willingness to voluntarily participate in the study and to provide written informed consent prior to enrollment.

Exclusion Criteria:

1. A confirmed previous diagnosis of other psychiatric disorders, including intellectual disability, bipolar disorder, treatment-resistant depression, or suicidal ideation.
2. Pregnant or breastfeeding women.
3. Individuals with known food or drug allergies, or those with alcohol abuse or psychotropic substance abuse.
4. Use of antibiotics or probiotics known to affect gut microbiota for more than one week within one month prior to enrollment.
5. Participants who withdrew from the study, discontinued intervention, or were unable to complete the study for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Assess the changes in the severity of depressive symptoms. | 8 weeks
  The severity of depressive symptoms is assessed by changes in scores on the Hamilton Depression Rating Scale-17 items (HAMD-17) and the Hamilton Anxiety Rating Scale (HAMA-14). The Hamilton Depression Rating Scale (17-item version) is a clinician-administered rating scale consisting of 17 items. The total score ranges from 0 to 52, with higher scores indicating more severe depressive symptoms. The Hamilton Anxiety Rating Scale (14-item version) is a clinician-administered rating scale consisting of 14 items. The total score ranges from 0 to 56, with higher scores indicating more severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan University of Science and Technolog, Luoyang, Henan, China